CLINICAL TRIAL: NCT03523793
Title: Health System Implementation of Clinical Practice Guidelines for Neck and Low Back Pain in Outpatient Physical Therapy Settings
Brief Title: Clinical Practice Guidelines for Neck and Low Back Pain in Outpatient Physical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Foundation for Physical Therapy Research (Other); Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201800569; 0045970 (710850-6) (Other: University of Pittsburgh); 00000775 (Other Grant/Funding Number: Foundation for Physical Therapy)
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain; Low Back Pain
Keywords: Outpatient Physical Therapy
MeSH Terms: conditions — Neck Pain; Low Back Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: cross-sectional stepped wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapists - CPG (Experimental): Cross-sectional stepped wedge design with 16 physical therapy clinics (including approximately 40 physical therapists) being allocated to one of 4 sequences that differ in CPG implementation time (each sequence consisting of 4 clinics). This proposed study will be conducted over 68 weeks, with the initial 12 weeks serving as a baseline washout phase (before any clinic has received training), then 4 clinics crossing over from standard care (control) to CPG and decision support tool implementation (intervention) approximately every 8 weeks until week 44 when all 4 sequences (16 clinics) have completed training.
  Interventions: Behavioral: Clinical Practice Guideline Implementation
- Physical Therapists - Control (Active Comparator): This proposed study will be conducted over 68 weeks, with the initial 12 weeks serving as a baseline washout phase (before any clinic has received training), then 4 clinics crossing over from standard care (control) to CPG and decision support tool implementation (intervention) approximately every 8 weeks until week 44 when all 4 sequences (16 clinics) have completed training.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Clinical Practice Guideline Implementation — The Study team will use several methods from the implementation strategy taxonomy of the Effective Practice and Organization of Care (EPOC) classification system to improve our likelihood for successful neck and low back pain implementation consisting of: 1) educational materials, workshops and outreach visits from trainers; 2) external consultant testimonials; 3) iterative quality improvement processes (including ongoing analysis of clinician feedback to improve process); 4) routine collection of patient reported outcomes to engage discussion among clinician groups and outpatient division leaders) and 5) local organization consensus process (including feedback from key outpatient division stakeholders).
  Arms: Physical Therapists - CPG
Other: Standard Care — Considering the stepped wedge design with a 12-week washout phase, clinics will be providing standard physical therapy prior to receiving clinical practice guideline training.
  Arms: Physical Therapists - Control

SUMMARY:
This study will investigate implementation of a process to enhance Clinical Practice Guideline (CPG) adherence to limit unwarranted variability in initial treatment decisions with high potential for providing more effective and efficient physical therapy management for patients with neck and low back pain.

DETAILED DESCRIPTION:
Effective implementation of CPGs to augment initial clinical decision making during physical therapy management of patients with spine related musculoskeletal pain will have several important goals: 1) improve patient pain and disability outcomes, 2) limit over utilization of physical therapy services, and 3) increase adherence to limit unwarranted variation in clinical practice. This proposed pilot study proposal will test if a multifaceted intervention strategy for implementation of neck and low back CPG meets these goals and provide necessary data for larger system wide implementation efforts.

Specific Aim 1: Determine if physical therapy clinics that receive neck and low back pain (LBP) clinical practice guideline (CPG) training are associated with improved patient outcomes compared to those that have not received training. Neck and LBP specific disability and pain intensity will be assessed at intake, on a weekly basis and at discharge (Specific Aim 1a). Secondary patient outcomes will consist of patient satisfaction scores (Specific Aim 1b). Statistical analyses will evaluate for temporal effects of training considering the stepped wedge study design.

Specific Aim 2: Determine if multifaceted interventions for CPG implementation positively impacts physical therapist beliefs, attitudes, knowledge and behaviors over time. CPG adherence (by clinicians) will be indirectly assessed using quantitative and qualitative methods consisting of: 1) clinician checklists, 2) clinician questionnaires, 3) quality indicators, and 4) total proportion outcome measure assessments (Specific Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Receiving outpatient physical therapy for a diagnosis covered in previously published CPGs for neck or LBP
* Able to read and comprehend English language (necessary for completion of self-report e-forms)

Exclusion Criteria:

* Any diagnosis indicating systemic involvement
* Widespread chronic pain syndrome
* Neuropathic pain syndromes
* Neurological disorders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1441 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 68 weeks
  The Oswestry Disability Index (ODI), which has 10 items that assesses how low back pain affects common daily activities. The ODI has a range of 0% "no disability due to low back pain" to 100% "completely disabled due to low back pain", with higher scores indicating higher disability from low back pain.
Neck Disability Index (NDI) | 68 weeks
  The Neck Disability Index (NDI), which has 10 items that assesses how neck pain affects common daily activities. The NDI has a range of 0% "no disability due to neck pain" to 100% "completely disabled due to neck pain", with higher scores indicating higher disability from neck pain.
Numeric Pain Rating Scale (NPRS) | 68 weeks
  Numeric Pain Rating Scale (NPRS) Pain intensity will be rated using a NPRS, ranging from "0" (no pain) to "10" (worst pain imaginable). Patients will be asked to rate their current pain intensity, as well as their best and worst level of pain intensity over the past 24 hours. These 3 pain ratings will averaged and used as the NPRS variable in this study.

SECONDARY OUTCOMES:
Rehabilitation Outpatient Division Patient Satisfaction Survey | 68 weeks
  To assess overall therapy experience and explanations provided by therapist.
Evidence-Based Practice Questionnaire (EBPQ) | 68 weeks
  The Evidence-Based Practice Questionnaire (EBPQ) to assess clinician beliefs, attitudes, knowledge and self-reported behaviors regarding evidence-based practice and clinical practice guidelines. Responses range from Strongly Agree to Strongly Disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Beneciuk, DPT,PhD,MPH, Principal Investigator — University of Florida; Brooks Rehabilitation
Locations (1):
- Brooks Rehabilitation, Jacksonville, Florida, United States

REFERENCES:
- [Background] Beneciuk JM, Osborne R, Hagist MB, Crittenden J, Buzzanca KE, Gao H, Wu SS. American Physical Therapy Association Clinical Practice Guideline Implementation for Neck and Low Back Pain in Outpatient Physical Therapy: A Nonrandomized, Cross-sectional Stepped-Wedge Pilot Study. J Orthop Sports Phys Ther. 2022 Feb;52(2):113-123. doi: 10.2519/jospt.2022.10545. PMID 35100820
- See also: Primary Results — https://pubmed.ncbi.nlm.nih.gov/35100820/